CLINICAL TRIAL: NCT04791332
Title: A Double-blind, Placebo-controlled, Randomized, Single Ascending and Multiple Dose Study to Investigate the Safety, Tolerability and Pharmacokinetics of JNJ-67953964 in Healthy Japanese Adult Male Participants
Brief Title: A Study of JNJ-67953964 in Healthy Japanese Adult Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR108983; 67953964EDI1002 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2021-03-09; First posted 2021-03-10 (Actual); Last update posted 2025-04-28 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Aticaprant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Dose Cohort: Cohort 1 and 2 (Experimental): Participants will receive a single oral dose of JNJ-67953964 or a matching placebo on Day 1.
  Interventions: Drug: JNJ-67953964; Drug: Placebo
- Multiple Dose Cohort: Cohort 3 (Experimental): Participants will receive multiple oral dose of JNJ-67953964 once daily or a matching placebo up to Day 14.
  Interventions: Drug: JNJ-67953964; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-67953964 — JNJ-67953964 capsule will be administered orally.
Drug: Placebo — Matching placebo will be administered orally.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) after single- and multiple-dose oral administration of JNJ-67953964 in healthy Japanese adult male participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be healthy on the basis of physical and neurological examination, medical history, vital signs, and 12- lead electrocardiogram (ECG) (QT corrected according to Fridericia's formula [QTcF] less than or equal to [<=] 450 milliseconds [msec]) performed at screening and admission to the clinical site. Minor abnormalities in ECG, which are not considered to be of clinical significance by the investigator, are acceptable. The presence of left bundle branch block, atrioventricular (AV) block (second degree or higher), or a permanent pacemaker or implantable cardioverter defibrillator will lead to exclusion
* Participant must be healthy on the basis of clinical laboratory tests performed at screening and baseline (Day -1). If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, retesting of an abnormal lab value(s) that may lead to exclusion will be allowed once during the screening phase upon discretion of the investigator. At screening and baseline (Day -1), alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase, and bilirubin must be within normal ranges. The participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study according to both the investigator and to the study responsible physician (SRP), are acceptable. This determination must be recorded in the participant's source documents and initialed by the investigator
* Body mass index (BMI; weight in kilogram divided by the square of height in meters between 18 and 30 kilogram per meter square (kg/m^2) (inclusive), and body weight not less than 50 kg at screening and on Day -1
* Men who are sexually active with a woman of childbearing potential and have not had a vasectomy must agree to use a barrier method of birth control example, a condom for the duration of the study plus 3 months after receiving the last dose of study intervention, and all men must not donate sperm during the study and for 3 months after receiving the last dose of study intervention. In addition, their female partners should also use an additional method of birth control (which may include a hormonal method, an intrauterine device [IUD] or an intrauterine system [IUS]) for at least the same duration
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 139 millimeters of mercury (mmHg) systolic, inclusive, and no higher than 89 mm Hg diastolic at screening and on Day -1. If blood pressure is out of range, up to 2 repeated assessments are permitted

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, lipid abnormalities, bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency thyroid disease, Parkinson's disease, infection including participants with a positive of severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) specific test on Day -8 to -1, or any other illness that the Investigator considers should exclude the participant
* Known allergies, hypersensitivity, or intolerance to JNJ-67953964 and its excipients
* History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5) criteria within 6 months before screening or positive test result(s) for alcohol, nicotine metabolites and/or drugs of abuse (opiates [including methadone], cocaine, amphetamines, methamphetamines, cannabinoids, barbiturates, ecstasy, and benzodiazepines) at screening or at admission to the study center
* History of clinically significant drug and/or food allergies
* Clinically significant acute illness within 7 days prior to study intervention administration

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) for Single- dose Cohort | Up to 5 weeks
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with AEs for Multiple- dose Cohort | Up to 7 weeks
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Plasma Concentration of JNJ-67953964 for Single- dose Cohort | Up to Day 5
  Plasma samples will be analyzed to determine concentrations of JNJ-67953964 using a fully validated liquid chromatography coupled to tandem mass spectrometry (LC-MS/MS) method.
Plasma Concentration of JNJ-67953964 for Multiple- dose Cohort | Up to Day 17
  Plasma samples will be analyzed to determine concentrations of JNJ-67953964 using a fully validated LC-MS/MS method.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Sumida Hospital, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency